CLINICAL TRIAL: NCT02410629
Title: Influence of Timing on Motor Learning
Brief Title: To Determine the Therapeutic Effect of the Music Glove and Conventional Hand Exercises to Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Reinkensmeyer (Other)
Responsible Party: Sponsor-Investigator, David Reinkensmeyer, Assistant Professor, Department of Neurology, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 2008-6432
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Glove (Experimental): Music Glove is a glove with sensors attached to the tips of all 5 fingers. The glove is connected to a software musical program like guitar hero. Participants will follow the rhythm or musical notes of the songs and move their fingers accordingly. Participants are reinforced with biofeedback that includes visual and auditory cues when the correct sequences are achieved.
  Interventions: Device: Music Glove
- Conventional Hand Exercise Program (Active Comparator): Conventional Hand Exercise Program includes range of motion exercises, strengthening exercises, coordinating exercises of the hand and fingers. This exercise program is designed by an occupational therapist and is a general exercise program that a stroke patient will receive when he/she is being discharged from the hospital.
  Interventions: Other: Conventional Hand Exercise Program

INTERVENTIONS:
Device: Music Glove — Participants will exercise at home using the music glove for 3 times a week for 3 weeks with a minimal of 3 hours per week.
  Arms: Music Glove
Other: Conventional Hand Exercise Program — Participants will exercise at home using the hand exercise program designed by an occupational therapist for 3 times a week for 3 weeks with a minimal of 3 hours per week.
  Arms: Conventional Hand Exercise Program

SUMMARY:
The investigators are trying to determine the therapeutic effect of the music glove and conventional hand exercise program to the subacute stroke patients. All participants will be randomized into two groups: AB and BA. They will all exercise at least 3 times a week for 3 weeks with a minimal 3 hours exercise time per week. Participants will receive the other intervention at 3-month post stroke date. Clinical evaluations will be performed at baseline, post therapy after first intervention, 3-week post intervention follow up, 3-month post stroke, post therapy after second intervention, 3-week post second intervention follow up, and 6-month post stroke follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* History of a single stroke at least 1 week prior to enrollment
* Upper Extremity weakness measured on a standard clinical scale
* No active major psychiatric problems, or neurological/orthopedic problems affecting the stroke affected upper extremity
* No active major neurological disease other than the stroke
* Absence of pain in the affected upper extremity

Exclusion Criteria:

* Severe tone at the affected upper extremity as measured on a standard clinical scale
* Severe aphasia as measured on a standard clinical scale
* Severe reduced level of consciousness
* Severe sensory/proprioception deficit at the affected upper extremity as measured on a standard clinical scale
* Currently pregnant
* Difficulty in understanding or complying with instructions given by the experimenter
* Inability to perform the experimental task that will be studied
* Increased pain with movement of the affected upper extremity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: An Do, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Music Glove First Then Conventional Hand Exercise Program: Music Glove is a glove with sensors attached to the tips of all 5 fingers. The glove is connected to a software musical program like guitar hero. Participants will follow the rhythm or musical notes of the songs and move their fingers accordingly. Participants are reinforced with biofeedback that includes visual and auditory cues when the correct sequences are achieved.
  Music Glove: Participants will exercise at home using the music glove for 3 times a week for 3 weeks with a minimal of 3 hours per week.
- Conventional Hand Exercise Program First Then Music Glove: Conventional Hand Exercise Program includes range of motion exercises, strengthening exercises, coordinating exercises of the hand and fingers. This exercise program is designed by an occupational therapist and is a general exercise program that a stroke patient will receive when he/she is being discharged from the hospital.
  Conventional Hand Exercise Program: Participants will exercise at home using the hand exercise program designed by an occupational therapist for 3 times a week for 3 weeks with a minimal of 3 hours per week.
Period: Overall Study
Arm/Group | Music Glove First Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First Then Music Glove
Started | 8 | 9
Completed | 5 (5 subjects from the music glove group were crossed over to conventional hand exercise group.) | 6 (6 subjects from the conventional hand exercise group were crossed over to music glove group.)
Not Completed | 3 | 3
Not completed — Family cannot commit to the study | 2 | 1
Not completed — Subject returned to work | 1 | 0
Not completed — Subject moved back to home country | 0 | 1
Not completed — Subject underwent heart surgery | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Music Glove First - Conventional Second: Music Glove is a glove with sensors attached to the tips of all 5 fingers. The glove is connected to a software musical program like guitar hero. Participants will follow the rhythm or musical notes of the songs and move their fingers accordingly. Participants are reinforced with biofeedback that includes visual and auditory cues when the correct sequences are achieved.
  Music Glove: Participants will exercise at home using the music glove for 3 times a week for 3 weeks with a minimal of 3 hours per week.
- Conventional Hand Exercise Program First - Music Glove Second: Conventional Hand Exercise Program includes range of motion exercises, strengthening exercises, coordinating exercises of the hand and fingers. This exercise program is designed by an occupational therapist and is a general exercise program that a stroke patient will receive when he/she is being discharged from the hospital.
  Conventional Hand Exercise Program: Participants will exercise at home using the hand exercise program designed by an occupational therapist for 3 times a week for 3 weeks with a minimal of 3 hours per week.
- Total: Total of all reporting groups
Arm/Group | Music Glove First - Conventional Second | Conventional Hand Exercise Program First - Music Glove Second | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (17) | 59 (13) | 62 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Box and Block Test
Description: We compared the change of Box and Block Test scores from baseline evaluation to the end of 3-week of therapy (Intervention 1), and from 12-week post-stroke to end of 3-week therapy (Intervention 2). Participants are instructed to move as many blocks as possible, one at a time, from one compartment in a box to a second compartment over a divider for a period of 60 seconds; each block that is moved is counted, and multiple blocks moved at the same time are counted as a single block. The higher scores indicates a better outcome.
Time Frame: From baseline to end of therapy (3 weeks)
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | Music Glove First Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First Then Music Glove
Number analyzed (Participants) | 6 | 5
blocks
  Baseline evaluation | 21 (14) | 33 (15)
  Change in Post therapy evaluation (Intervention 1) | 12 (4) | 7 (5)
  Change in 16-week post cross over evaluation | 19 (16) | 12 (11)

2. Secondary Outcome: Fugl-Meyer Motor Assessment of the Upper Extremity
Description: We measure the change of the Fugl-Meyer Motor Assessment scores from the baseline evaluation to 3-week therapy (intervention 1) and 12-week post-stroke to end of 3-week therapy (Intervention 2). Fugl-Meyer is a 66-point scale measuring the movement pattern of upper extremities. For this study, we analyze total score only. The higher scores indicate a better outcome.
Time Frame: From baseline to end of therapy (3 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Music Glove First Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First Then Music Glove
Number analyzed (Participants) | 6 | 5
scores on a scale
  Baseline evaluation | 44 (13) | 42 (9)
  Change in Post therapy evaluation | 4 (5) | 7 (11)
  Change in 16-week post cross over evaluation | 9 (8) | 9 (10)

3. Secondary Outcome: Action Research Arm Test
Description: We compared the change in Action Research Arm Test (ARAT) scores from the baseline evaluation to 3-week therapy (Intervention 1) and 12-week post-stroke to 3-week therapy (Intervention 2). The ARAT is a 57-point scale which measures upper extremity function, coordination, and dexterity. The higher scores indicate a better outcome.
Time Frame: From baseline to end of therapy (3 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Music Glove First Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First Then Music Glove
Number analyzed (Participants) | 6 | 5
scores on a scale
  Baseline evaluation | 42 (14) | 47 (12)
  Change in Post therapy evaluation | 9 (9) | 7 (13)
  Change in 16-week post cross over evaluation | 13 (14) | 7 (13)

4. Secondary Outcome: 9-Hole Peg Test
Description: We compared the change in 9-Hole Peg Test scores from the baseline evaluation to 3-week therapy (Intervention 1) and 12-week post-stroke to 3-week therapy (Intervention 2). The 9-Hole Peg Test is a timed test that measures the time it takes to place, and remove 9 pegs. The maximum allowed time for the test is 60 seconds. The more number of pegs placed and removed indicate a better outcome. The shorter time it takes to complete the task indicates a better outcome.
Time Frame: From baseline to end of therapy (3 week)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Music Glove First Then Conventional Hand Exercise Program | Conventional Hand Exercise Program First Then Music Glove
Number analyzed (Participants) | 6 | 5
seconds
  Baseline 9-Hole Peg Test Scores | 55 (12) | 47 (15)
  Change in post therapy score (Intervention 1) | -5 (8) | -7 (4)
  Change in 16-week post cross over evaluation | -9 (12) | -5 (8)

ADVERSE EVENTS:
Arm/Group | Music Glove First - Conventional Second | Conventional Hand Exercise Program First - Music Glove Second
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No